CLINICAL TRIAL: NCT03100071
Title: A Pilot Study in Cancer Patients With Central Venous Catheter (CVC) Associated Deep Vein Thrombosis (DVT) in the Upper Extremity Treated With Low Molecular Weight Heparin (LMWH) and Apixaban (Catheter 3)
Brief Title: Central Venous Catheter (CVC) Associated Deep Vein Thrombosis (DVT) in Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Michael Kovacs (Other)
Collaborators: Ottawa Hospital Research Institute (Other); Jewish General Hospital (Other)
Responsible Party: Sponsor-Investigator, Michael Kovacs, Associate Professor, Medical Doctor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: R-17-160
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Cancer Patients; Central Venous Catheter Thrombosis; Upper Extremity Thrombosis
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis | interventions — apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Apixaban — Patients will be treated with Low Molecular Weight Heparin (LMWH) for 1 week and then with apixaban 5 milligram (mg) twice daily for 11 weeks.
  Other Names: Eliquis

SUMMARY:
Cancer patients with Central Venous Catheter (CVC) Associated Deep Vein Thrombosis (DVT) will be treated with Low Molecular Weight Heparin (LMWH) and apixaban. Study duration is 12 weeks.

DETAILED DESCRIPTION:
Cancer patients who have developed blood clot in the arm that has the central venous catheter will be treated with standard of care blood thinning injection of low molecular weight heparin for 1 week and then for apixaban 5 mg twice daily for the rest of 11 weeks. Data will be collected to see if the central venous catheter "survived" or remained in place and did not have to be taken out because of the clot.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age.
2. Symptomatic acute upper limb thrombosis in the axillary, subclavian or internal jugular veins, with or without pulmonary embolism, associated with central venous catheter objectively documented by compression ultrasonography, venogram or Computerized Tomography (CT) scan.
3. Diagnosis of active malignancy, as defined by patients who are either receiving active treatment, or have metastatic disease or who have been diagnosed within the past two years.
4. Willing to provide written informed consent.

Exclusion Criteria:

1. Presence of dialysis catheters
2. Active bleeding or high risk for major bleeding
3. Platelet Count < 75 x 109/L
4. Creatinine Clearance < 30 mL/min
5. Currently on other anticoagulant with therapeutic intent for another indication
6. Pulmonary embolism accompanied by hemodynamic instability or oxygen requirement
7. Inability to infuse through the catheter after a trial of intraluminal thrombolytic therapy (2 mg tPA).
8. Patients with Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL) or multiple myeloma with a bone marrow or stem cell transplant planned within the next 3 months
9. Treatment for current episode > 7 days with any acceptable anticoagulant therapy
10. Concomitant use of p-glucoprotein and Cytochrome P450 3A4 (CYP3A4) inhibitors (for example azole antifungals such as ketoconazole) or inducers (for example rifampicin, antiepileptics)
11. Recent coronary artery stent requiring dual anti-platelet therapy (for example acetylsalicylic acid [ASA] and Plavix)
12. If female of childbearing potential: pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer patients with central venous catheter associated deep vein thrombosis in the upper extremity
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Central Line Failure | within 3 months of study follow-up
  Infusion failure that does not respond to 2 milligram (mg) tissue Plasminogen Activator (tPA)

SECONDARY OUTCOMES:
Recurrent Venous Thromboembolism (VTE) | within 3 months of study follow-up
  recurrence of blood clot either in leg or lung or both
Bleeding | within 3 months of study follow-up
  Major bleeding, clinically relevant minor bleed, death, time to central line failure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kovacs, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (2):
- Canada (2):
  - London Health Science Center, Victoria Hospital, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No